CLINICAL TRIAL: NCT04755725
Title: Comparison Between Epidural Catheter and Surgically Implanted Rectus Sheath Catheter in Management of Postoperative Pain Following Laparotomy
Brief Title: Epidural Catheter and Surgically Implanted Rectus Sheath Catheter in Management of Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, rabab Mohammad habeeb, principal investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5/2017ANET
Record Dates: First submitted 2021-02-03; First posted 2021-02-16 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Pain
Keywords: rectus sheath catheter, pain following laparotomys.
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural Group (Active Comparator): epidural catheter inserted pre induction
  Interventions: Device: Epidural catheter
- Rectus sheath catheter Group (Active Comparator): rectus sheath catheter inserted by the surgeon at the end of surgery
  Interventions: Device: rectus sheath catheter

INTERVENTIONS:
Device: Epidural catheter — epidural catheter inserted pre induction
  Arms: Epidural Group
Device: rectus sheath catheter — The surgeon will place one hand inside the abdomen and with the other hand inserted the Tuohy needle through the skin and fascia. The surgeon will feel when the needle tip is just superfacial to interface between the peritoneum and muscle layer and avoid penetration of inferior epigastric artery. The procedure will be repeated on the contralateral
  Arms: Rectus sheath catheter Group

SUMMARY:
One hundred and twenty patients at age range from 18 to 60 undergoing laparotomy was enrolled in this study. Patients were randomly assigned to two groups 60 in epidural group and the other 60 patients in rectus catheter group. epidural catheter inserted pre induction but rectus sheath catheter inserted by the surgeon at the end of surgery.

DETAILED DESCRIPTION:
One hundred and twenty patients at age range from 18 to 60 undergoing laparotomy was enrolled in this study. Patients were randomly assigned to two groups 60 in epidural group and the other 60 patients in rectus catheter group. epidural catheter inserted pre induction but rectus sheath catheter inserted by the surgeon at the end of surgery. In both groups we activated with10 ml bupivacain25% before patient recovery then 10 ml bupivacain.125% each 6 hours. If patient still in pain 1gm perflgan injected. If patient still in pain 10 mg nalufine for 70 kg patient injected. we will record pulse, blood pressure and visual analogue scale at 0,6,12,24 and 36 hours postoperative. Also Occurrence of nausea and vomiting, Time of return of bowel movement, Time of discharage and amount of analgesia used will be recorded. Results, discution will be later.

ELIGIBILITY:
Inclusion Criteria:

* patients at age rang from 18 to 60 undergoing laparotomy
* patients ASA1,2 physical status

Exclusion Criteria:

* any known coagulopathy
* morbid obesity
* kyphosis or scoliosis
* those with known sensitivity to local anesthetic drugs
* lack of cooperation and inability to understand or perform verbal or physical assessments.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain relief | 36hours
  Measured by Visual Analogue Scale (VAS) pain measurement scale divided from 0 to 10 where 0 is no pain and10 worst pain can be imagined

SECONDARY OUTCOMES:
Side effects | 36hours
  Occurrence any side effects Time of return of bowel movement. Time of discharage. Amount of analgesia used
Total of analgesic consumption | 36 hours
  total consumption of naluphine and paracetamol pre milligram

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Raouf, Professor, Study Chair — Menoufia University
Locations (2):
- Egypt (2):
  - Faculty of Medicine Menoufia University, Cairo, Governorate
  - Menoufia University, Cairo, Governorate

IPD SHARING:
Plan to Share IPD: No